CLINICAL TRIAL: NCT05472454
Title: The Ready-to-EAt Meals for Cardiovascular Health (REACH) Study
Brief Title: The Ready-to-Eat Meals for Cardiovascular Health Study
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Pablo Monsivais, Associate Professor, Washington State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19288-001
Record Dates: First submitted 2022-07-15; First posted 2022-07-25 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Diet; Hypertension; Cardiovascular Diseases; Blood Pressure
Keywords: DASH; Dietary Approaches to Stop Hypertension; Meals; High Blood Pressure; Hypertension
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — Fast Foods

STUDY DESIGN:
Intervention Model Description: Pre-post design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ready-to-eat meals (Other): Pre-Post
  Interventions: Other: Ready-to-eat meals

INTERVENTIONS:
Other: Ready-to-eat meals — Participant group to consume ready-to-eat meals in accordance with the DASH diet for a period of 4 weeks.

SUMMARY:
The proposed project explores the acceptability and health benefits of ready-to-eat (RTE) meals based on the Dietary Approaches to Stop Hypertension (DASH) eating plan. The researchers have developed 14 recipes following the DASH eating plan, which is recommended for the prevention of cardiovascular disease (CVD). The prepackaged meals will be processed using Washington State University (WSU) microwave technologies to ensure food safety. In this pilot study, a sample of 30 participants will be recruited by to study the impact of the DASH meals on blood pressure. All meals will be provided to participants, who will consume the meals daily over a period of 4 weeks. Daily and weekly monitoring of participants (blood pressure and weight) will allow us to gain a scientific understanding on the preventive power of healthy diets in lowering blood pressure and reducing CVD risk.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 years old or older
* BMI 18.5-40.0 kg/m2
* Daily access to working internet, microwave, refrigerator, and freezer
* English fluency

Exclusion Criteria:

* Regular use of drugs that affect BP, including weight loss medications
* Diagnosed hypertension OR systolic BP >130 and/or diastolic BP >80
* Diagnosis of any hypotensive disorders OR systolic BP <100 and/or diastolic BP<65
* Dietary restrictions, including allergy/intolerances
* Presence or history of diabetes
* Previous cardiac event, congestive heart failure, or angina
* Weight loss or gain>15lb in previous 3 months
* Following a diet to increase or decrease body weight
* Cancer diagnosis or treatment in past 2 years
* ≥14 alcoholic drinks/week for men; ≥ 7 alcoholic drinks/week for women
* Use of nicotine, marijuana, or illicit drugs
* Pregnancy, planned pregnancy, or breastfeeding
* Inability to comprehend the nature of the study or instructions
* No access to the internet
* Planning to leave the Spokane area during the study
* Not fluent in the English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure | through study completion, measured weekly for 5 weeks
  To determine dietary patterns on blood pressure using an omron blood pressure monitor.

SECONDARY OUTCOMES:
Body weight (kg) | through study completion, measured weekly for 5 weeks
  To determine dietary patterns on body weight (kg) using a Angel USA 400 Pound Physician Digital Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Monsivais, PhD, MPH, Principal Investigator — Washington State University
Locations (1):
- Washington State University, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No